CLINICAL TRIAL: NCT04091100
Title: Effects of Electroacupuncture and Myofascial Release on Pain, Neck Functions and Depression Status in Patients With Tension-Type Headaches
Brief Title: Effects of Electroacupuncture and Myofascial Release on Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Leyla Ataş Balcı, Assist. Prof, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAB2
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Tension-Type Headache
Keywords: Pain; Acupuncture; Tension-Type Headache; Myofascial Releasing; Depression
MeSH Terms: conditions — Tension-Type Headache; Pain; Depression | interventions — Electroacupuncture; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: The individuals were randomly allocated into electroacupuncture and myofascial release groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Active Comparator): The individuals in the electroacupuncture group were administered the therapy by a certified acupuncturist. Two Shenlong acupuncture needles were inserted in each of the trapezius and levator scapulae muscles at intervals of 0-3 mm and clips were attached to their ends. Afterwards, an electrical current of 2 mA and 60 Hz was administered using the Enraf Nonius Sonoplus 492 (OPTOMED) device for 20 minutes.
  Interventions: Procedure: Electroacupuncture
- myofascial release (Active Comparator): Firstly, longitudinal stretching was done with forearm to the muscles in the person's neck in order to relax. Afterwards, the researcher placed one hand under the person's head and placed their fingertips on the muscles under the occipital bone in the neck area. The researcher applied lateral flexion to the neck with one hand while placing the other hand on the trapezius and levator scapulae muscles and then stretched the muscles with friction massage. After this step, the participant's neck was guided back into a neutral position and the pinching technique was applied to the muscles. During the administration of therapies, the trigger points on muscles were identified and friction was applied to these sites until a loosening could be felt. The myofascial release sessions concluded with the administration of the friction massage technique once again to the muscles.
  Interventions: Procedure: Myofascial Release

INTERVENTIONS:
Procedure: Electroacupuncture — An electrical current of 2 mA and 60 Hz was administered using the Enraf Nonius Sonoplus 492 (OPTOMED) device for 20 minutes. All the treatments were performed for 2 sessions per week for 3 weeks. Both groups were given a home program involving neck stretching and posture exercises. The exercises were to be performed at least two times a day in two sets of fifteen repetitions.
  Arms: electroacupuncture
Procedure: Myofascial Release — longitudinal stretching, friction massage and pinching technique, All the treatments were performed for 2 sessions per week for 3 weeks. Both groups were given a home program involving neck stretching and posture exercises. The exercises were to be performed at least two times a day in two sets of fifteen repetitions.
  Arms: myofascial release

SUMMARY:
Tension-type headaches (TTH) last from thirty minutes to seven days, were ranked second among the primary types of headaches. The diagnosis of TTH is made according to the diagnostic criteria of the Second Beta version of the International Classification of Headache Disorders. The causes of TTH include the activation of extremely tense peripheric afferent neurons through the head and neck muscles, muscle sensitivity and stress. Additionally, a limited range of motion (ROM) in the neck may also lead to TTH.

The treatment of TTH involve both pharmacological and non-pharmacological methods. It is known that the pharmacological treatment of TTH has a limited effect. However, previous studies have shown that physical therapy programs that include methods such as acupuncture, Transcutaneous Electrical Nerve Stimulation (TENS), exercise, biofeedback, manipulation, cryotherapy, massage, strengthening of the neck muscles, stretching exercises are effective in alleviating TTH.

It has been observed that the trigger points in muscles play a role in TTH. Trigger points are generally defined as hyper-irritable points inside taut bands. It has been demonstrated that myofascial release, which is applied to the trigger points and is effective in relaxation treatments through stimulation of the neuromuscular system, relieves headaches via muscle relaxation. Electroacupuncture is another method used in relieving myofascial pain origin that involves the application of acupuncture needles to particular points and delivery of an electrical current at a specific frequency. The stimulation of muscle and skin tissues in affected areas is carried out by means of needles and the electrical current relieves pain and muscle spasms. In a meta-analysis study, it was found that electroacupuncture had a higher pain-relieving effect. However, a review of related studies deemed them to be lacking because the assessments were too limited to make it possible to unequivocally state that electroacupuncture has a high level of therapeutic efficacy.

The studies performed, however, did not examine the efficacy of electroacupuncture and myofascial release on TTH. Given that situation, the purpose of our study is to investigate the effects of electroacupuncture and myofascial release applied to points of tension in the neck muscles and trigger points of people suffering from TTH in terms of the headache intensity and frequency, neck functions, sleep quality and depression status.

DETAILED DESCRIPTION:
The 19 individuals who were referred to Bahçeşehir University's Department of Physiotherapy and Rehabilitation at the School of Health Sciences, with TTH, and who were 18 years of age and older, were recruited for the study. The individuals were randomly allocated into electroacupuncture and myofascial release groups with the Research Randomizer program.

Evaluation Methods A Visual Analogue Scale (VAS) to evaluate pain levels of the participants, CROM (Cervical Range of Motion) to evaluate neck ROM, Beck's Depression Inventory to evaluate depression status, Neck Pain Disability Scale to evaluate to evaluate the effect of their neck pain on the activities of the daily living Headache Diary to evaluate clinical features of the headache

ELIGIBILITY:
Inclusion Criteria:

* Indiviuals with cervical tension headache
* aged 18 years or older
* Accepting voluntary participation in the study

Exclusion Criteria:

* Epilepsy seizures,
* Heart disease
* Pacemaker,
* Patients with a history of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity at Three Weeks | 3 weeks
  VAS, is used to evaluate the intensity of pain, using a scale comprised of a 100-mm-long horizontal line and ending with at both ends by descriptors of pain intensity beginning with "no pain" to "extreme pain. Patients are asked to indicate their levels of pain on this range by placing a dot on the line
Change from Baseline Headache Intensity at Three Weeks | 3 weeks
  Headache diary (HD): Patients kept an HD for three weeks to record the clinical features of their headaches. In this diary, subjects documented the number of days per week that they experienced a headache, the duration of each headache (hour/day), and the headache intensity on a 5-point numerical pain rating scale (0: no pain, 5: maximum pain). For each subject, Headache index (HI) was calculated for the first and last ten days of the intervention period as following:
  Headache index (HI) = mean headache intensity X mean number of days with headache X mean duration of headache
Change from Baseline Range of Motion of the Neck at Three Weeks | 3 weeks
  The join ROM of the neck was measured via C-ROM goniometer which consists of two inclinometers for gravity on the sagittal and frontal planes, an inclinometer with magnetic needles that is inserted from above on the horizontal plane, a magnetic cervical collar, an arm with a ruler in cm units and a vertebral fixating arm with a balance system. This device has a plastic frame with a shape that is similar to a pair of glasses, as it rests on the nose and ears. During all measurements, the subjects were asked to sit on a chair with their arms held close to their bodies. Subjects were asked to look forward in a comfortable sitting position for the performance of the measurements. The initial position of each movement was set an angle of 0 degrees. The measurements were conducted while the subjects performed forward/backward bending, left/right side-bending and rotation movements on the left and right sides of the neck.
Change from Baseline Depression Status at Three Weeks | 3 weeks
  The Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory, which was developed to measure depression symptoms in adult individuals. The individuals assigned a score of 0 to 3 for the items of the 21-item scale, which measures characteristic attitudes and depression symptoms. The highest score that can be obtained on the scale is 63, while the threshold value is considered to be 17.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla ATAŞ BALCI, Principal Investigator — Bahçeşehir University, Department of Physiotherapy and Rehabilitation
Locations (1):
- Bahçeşehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chowdhury D. Tension type headache. Ann Indian Acad Neurol. 2012 Aug;15(Suppl 1):S83-8. doi: 10.4103/0972-2327.100023. PMID 23024570
- [Background] Karadaş, Ö. (2013) Gerilim Tipi Baş Ağrısı: Kronik Tip Değerlendirmesi, J Clin Anal Med, 4 (6), 522-6
- [Background] Madsen BK, Sogaard K, Andersen LL, Skotte J, Tornoe B, Jensen RH. Neck/shoulder function in tension-type headache patients and the effect of strength training. J Pain Res. 2018 Feb 23;11:445-454. doi: 10.2147/JPR.S146050. eCollection 2018. PMID 29503581
- [Background] Bendtsen L. Drug and Nondrug Treatment in Tension-type Headache. Ther Adv Neurol Disord. 2009 May;2(3):155-61. doi: 10.1177/1756285609102328. PMID 21179525
- [Background] Barbanti P, Egeo G, Aurilia C, Fofi L. Treatment of tension-type headache: from old myths to modern concepts. Neurol Sci. 2014 May;35 Suppl 1:17-21. doi: 10.1007/s10072-014-1735-3. PMID 24867829
- [Background] Georgoudis G, Felah B, Nikolaidis PT, Papandreou M, Mitsiokappa E, Mavrogenis AF, Rosemann T, Knechtle B. The effect of physiotherapy and acupuncture on psychocognitive, somatic, quality of life, and disability characteristics in TTH patients. J Pain Res. 2018 Oct 23;11:2527-2535. doi: 10.2147/JPR.S178110. eCollection 2018. PMID 30425565
- [Background] Alonso-Blanco C, de-la-Llave-Rincon AI, Fernandez-de-las-Penas C. Muscle trigger point therapy in tension-type headache. Expert Rev Neurother. 2012 Mar;12(3):315-22. doi: 10.1586/ern.11.138. PMID 22364330
- [Background] McKenney K, Elder AS, Elder C, Hutchins A. Myofascial release as a treatment for orthopaedic conditions: a systematic review. J Athl Train. 2013 Jul-Aug;48(4):522-7. doi: 10.4085/1062-6050-48.3.17. Epub 2013 Apr 3. PMID 23725488
- [Background] Ulett GA, Han S, Han JS. Electroacupuncture: mechanisms and clinical application. Biol Psychiatry. 1998 Jul 15;44(2):129-38. doi: 10.1016/s0006-3223(97)00394-6. PMID 9646895
- [Background] Wu, B., Zhan, G., Lin, Lian, Q. (2017), Electroacupuncture for treatment of cervicogenic headache: A meta-analysis. Transl Perioper & Pain Med, 2 (2).
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Cheng LL, Ding MX, Xiong C, Zhou MY, Qiu ZY, Wang Q. Effects of electroacupuncture of different frequencies on the release profile of endogenous opioid peptides in the central nerve system of goats. Evid Based Complement Alternat Med. 2012;2012:476457. doi: 10.1155/2012/476457. Epub 2012 Oct 24. PMID 23133494
- [Background] Ajimsha MS. Effectiveness of direct vs indirect technique myofascial release in the management of tension-type headache. J Bodyw Mov Ther. 2011 Oct;15(4):431-5. doi: 10.1016/j.jbmt.2011.01.021. Epub 2011 Feb 11. PMID 21943616
- [Background] Melchart D, Streng A, Hoppe A, Brinkhaus B, Witt C, Wagenpfeil S, Pfaffenrath V, Hammes M, Hummelsberger J, Irnich D, Weidenhammer W, Willich SN, Linde K. Acupuncture in patients with tension-type headache: randomised controlled trial. BMJ. 2005 Aug 13;331(7513):376-82. doi: 10.1136/bmj.38512.405440.8F. Epub 2005 Jul 29. PMID 16055451
- [Background] Doraisamy, M. A., Kumar, C. P., & Gnanamuthu, C. (2010). Chronic tension type headache and the impact of myofascial trigger point release in the short term relief of headache. Global Journal of Health Science, 2(2), 238